# INFORMED CONSENT FORM

## Title of Study:

Effects of Meal Energy Density on Anthropometric Measurements, Some Metabolic Parameters, and Subjective Appetite in Women

#### **NCT Number:**

(Not yet assigned – to be updated upon registration)

#### **Document Date:**

November 1, 2023

## **Principal Investigator:**

Dr. Melike Nur EROGLU

Sakarya University of Applied Sciences

Email: melikeeroglu@subu.edu.tr

Phone: +90 5384982024

### **Co-Investigators:**

Dr. Beril Köse

Dr. Nomingerel Tseveldorj Dr. Büşra Sabur Öztürk

This document provides information about the clinical study mentioned above. Your participation is entirely voluntary. Please read this form carefully before deciding to take part.

#### 1. Introduction

You are being invited to participate in a research study. This document provides you with information about the study. Please read it carefully and feel free to ask any questions. Your participation is voluntary.

## 2. Purpose of the Study

The purpose of this study is to evaluate the effects of consuming half of the daily energy intake at breakfast versus dinner on body measurements, metabolic markers, and appetite levels in overweight or obese premenopausal women.

## 3. Study Procedures

- You will be randomly assigned to one of two diet plans:
- Breakfast Group (BG): 50% of daily energy at breakfast, 35% at lunch, 15% at dinner.
- Dinner Group (DG): 15% of daily energy at breakfast, 35% at lunch, 50% at dinner.
- The intervention period is 6 weeks.
- Measurements will be taken at baseline, week 3, and week 6.
- Blood samples will be collected before and after the study.
- Appetite will be assessed using visual analog scales.
- You will be asked to maintain your normal physical activity and complete food diaries weekly.

#### 4. Risks and Discomforts

- Minimal discomfort from blood sampling (e.g., bruising or soreness).
- Possible mild hunger or satiety effects due to dietary timing.

#### 5. Benefits

- You may gain insights into your eating habits and metabolic health.
- Results may contribute to scientific knowledge on diet timing and obesity management.

#### 6. Confidentiality

All your personal information and results will be kept confidential and used only for research purposes. Data will be stored securely and anonymized for analysis.

## 7. Voluntary Participation

Your participation is voluntary. You may refuse to participate or withdraw at any time without penalty or loss of benefits.

#### 8. Contact Information

If you have any questions about the study, you may contact:

- Principal Investigator: Dr. Büşra Sabur Öztürk

Email: busra.sabur12@gmail.com

Phone: +90 554 887 9463

## 9. Consent

| I have read and understood the information above. I voluntarily agree to participate in the | is |
|---|---|
| study. | |

| Participant's Name: | |
|---------------------------|-------|
| Participant's Signature: | <br>_ |
| Date: | |
| Investigator's Name: | <br>_ |
| Investigator's Signature: | <br> |
| Date: | |